CLINICAL TRIAL: NCT06168032
Title: Efficacy of COVID-19 Booster-Dose Vaccine for Re-infection Precaution and Dynamics of Specific Serum Antibodies in the Management of Lung Cancer Patients With Systemic Anti-cancer Treatment
Brief Title: COVID-19 Vaccine Effectiveness Against Recurrent Infection Among Lung Cancer Patients and Biomarker Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K4846
Record Dates: First submitted 2023-12-11; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 Recurrent; Lung Cancer; Vaccination; Antibody; Chemotherapy; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccinated group (Experimental): Any booster doses(without limitations in the subtypes or brands of the vaccines) recommended or approved by Chinese government will be administered once in the 6th months after latest confirmed COVID-19 infection and during the following 6 months, any conditions including repeated COVID19 infection, critical and/or severe conditions and all-cause death will be recorded.
  Interventions: Biological: Any Chinese government-recommended COVID-19 booster vaccine
- Non-vaccinated group (No Intervention): Patients unwilling to get vaccination will be allocated into these group, but any events including recurrent COVID19 infection, critical and/or severe conditions and all-cause death will be recorded in the following six months.

INTERVENTIONS:
Biological: Any Chinese government-recommended COVID-19 booster vaccine — Any Chinese government-recommended COVID-19 booster vaccine(such as Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine(Sf9 Cell) and so on) will be once administered in the sixth month after COVID19 infection.
  Arms: Vaccinated group

SUMMARY:
A prospective, open-label and parallel non-randomized control trial and biomarker research study is intended to compare incidence of repeated COVID-19 infection, severe pneumonitis and mortality between lung cancer patients undergoing systemic antitumor therapies who get vaccinated with 1 booster dose(majorly against XBB) and those who refuse. Meanwhile, a biomarker research is designed to monitor serum level dynamics of specific antibodies against COVID-19,analyze its correlation with incidence of breakthrough infection and further explore optimal periods for vaccination.

DETAILED DESCRIPTION:
A single booster dose will be administered depending on patients' willingness in the sixth month after symptomatic COVID-19 infection and status including repeated COVID19 infection, critical and/or severe conditions and all-cause death will be recorded during the next 6 months after vaccination or not. For antibody analysis, 5 ml blood samples will be collected from all of the included patients respectively in the 3rd ,4.5th and 6th months after latest occurrence of symptomatic infection and at the same timepoints after booster dose vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who agree to participate in the trial and sign the informed consents.
2. Male or female, ≥18 years old.
3. Diagnosed of lung carcinoma by histological and cytological examinations.
4. Undergoing systemic anti-tumor treatments including chemotherapy, immunotherapy, chemoimmunotherapy and targeted therapy.
5. Recorded history of COVID19 infection.
6. Sufficiently functional organs.
7. Eastern Cooperative Oncology Group performance score (PS) ranging from 0 to 2.

Exclusion Criteria:

1. Life expectance less than 3 months.
2. Less than 3 months since last confirmed COVID-19 infection.
3. Patients unable to return the hospital for follow-up.
4. Patients allergic to COVID-19 vaccine.
5. Patients with histories of severe treatment-related adverse events graded 3rd or higher, including those caused by antitumor therapies or immunization except recoverable granulocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1224 (Estimated)
Dates: Start 2023-12-08 (Estimated); Primary Completion 2026-12-08 (Estimated); Study Completion 2026-12-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of recurrent symptomatic COVID-19 infection among lung cancer patients treated with systemic antitumor therapies who get vaccinated 6 months after COVID-19 infection. | up to 8 weeks
  The incidence of any of the following events: confirmed COVID 19 infection by antigen test or PCR test, with at least one related symptom including fever, cough, expectoration, dyspnea, headache, diarrhea and so on.

SECONDARY OUTCOMES:
Incidence of critical and/or severe symptomatic COVID-19 infection among lung cancer patients treated with systemic antitumor therapies who get vaccinated 6 months after COVID-19 infection. | up to 8 weeks
  The incidence of the following events: COVID 19 infection confirmed by antigen test or PCR test and diagnosed of critical and/or severe pneumonitis.
All-cause mortality rate | up to 8 weeks
  The proportions of patients who died from any causes after enrollment.
Overall survival | up to 8 weeks
  The time length from enrollment to death from any causes.
Incidence of antitumor drug-related adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | up to 8 weeks
  Evaluate adverse events of any cause(except cancer-related events), treatment-related adverse events, immune-mediated adverse events according to NCI-CTCAE V5.0.
Incidence of adverse events following immunization | up to 8 weeks
  Evaluate immunization-related adverse events including local or systemic symptoms(excluding those caused by cancer or anti-canter treatments like chemotherapies, tyrosine kinase inhibitors, immune checkpoint inhibitors and so on）

OTHER OUTCOMES:
Exploratory biomarker analysis | up to 8 weeks
  5 ml blood samples will be collected in the 3rd ,4.5th and 6th months after symptomatic infection and at the same timepoints after booster dose vaccination(the interventional group) or of the successive 6 months(control group) to monitor the titre of specific sero-antibodies against COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The result of the study and all the supporting information will be shared in the form of published article.